CLINICAL TRIAL: NCT02980575
Title: Does Music During Pulmonary Rehabilitation in Individuals With Chronic Obstructive Pulmonary Disease (COPD) Improve Outcome? A Randomized Controlled Trial
Brief Title: Music During Pulmonary Rehabilitation for Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Respirologist, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-016-WP
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Music; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Music Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise with music (Experimental): Participants will listen to music when they exercise
  Interventions: Other: Music; Other: Exercise
- Exercise (Active Comparator): Participants will not listen to music when they exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Music
  Arms: Exercise with music
Other: Exercise

SUMMARY:
This study is aimed at determining whether listening to music during exercise will improve health-related outcomes for individuals with chronic obstructive pulmonary disease (COPD). Half of the participants will listen to music while they exercise and half will not listen to music. The study will follow participants during their pulmonary rehabilitation program and for 6 months following completion of the program.

DETAILED DESCRIPTION:
People with chronic obstructive pulmonary disease (COPD) are encouraged to undertake exercise training as part of their treatment. However, they often find themselves limited by breathlessness and tiredness in their legs. These barriers limit how much a person may benefit from an exercise program and how well they may keep up with a recommended schedule of exercise at home. One way of reducing feelings of breathlessness and leg tiredness is by listening to music during exercise.

The impact of adding music to exercise versus exercise alone has not been explored in the setting of pulmonary rehabilitation. This study is aimed at determining the effect of listening to music during exercise sessions on exercise capacity, symptom severity, quality of life and motivation to exercise.

People with COPD will be randomly allocated to exercise plus music or exercise alone. A music therapist will aid with music selection for the exercise plus music group and the music will be loaded onto a portable device that participants will listen to with earbuds. All participants will complete assessments before starting a pulmonary rehabilitation program, at the end of the 8-10 week program and 6 months following completion of the program. They will complete walking tests, report symptom severity and complete a series of questionnaires asking about their quality of life, symptoms and keenness to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD (physician diagnosis and spirometry with FEV1/FVC ratio <70) and smoking history of greater than 10 pack years
* Stable clinical state, with no acute exacerbations over the last 6 weeks
* Referred to pulmonary rehabilitation program

Exclusion Criteria:

* Predominant diagnosis other than COPD (asthma, bronchiectasis, interstitial lung disease)
* Co-morbidities (orthopaedic, neurological, cardiac) which might prevent safe exercise training
* Substantial hearing difficulties (inability to hear music adequately)
* Regularly uses music when exercising

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in end 6-minute walk test dyspnea and fatigue levels | Change from baseline to end of 8-week PR program or 6 month follow-up
  End test dyspnea and fatigue levels from best 6MWT
Multidimensional dyspnea profile | Change from baseline to end of 8-week PR program or 6 months follow-up

SECONDARY OUTCOMES:
Change in chronic respiratory disease questionnaire scores | Change from baseline to end of 8-week PR program or 6 month follow-up
Change in hospital anxiety and depression scale score | Change from baseline to end of 8-week PR program or 6 month follow-up
Change in multidimensional fatigue inventory score | Change from baseline to end of 8-week PR program or 6 month follow-up
Change in physical activity enjoyment scale score | Change from baseline to end of 8-week PR program or 6 month follow-up
Change in StepWatch physical acitvity monitor results | Change from baseline to end of 8-week PR program or 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Craigiburn Community Health Centre, Craigieburn, Victoria, Australia
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee AL, Butler SJ, Jung P, Clark IN, Tamplin J, Goldstein RS, Brooks D. Participant-selected music listening during pulmonary rehabilitation in people with chronic obstructive pulmonary disease: A randomised controlled trial. Chron Respir Dis. 2024 Jan-Dec;21:14799731241291065. doi: 10.1177/14799731241291065. PMID 39367818